CLINICAL TRIAL: NCT02704013
Title: Role of Urinary Neurotrophin and Cytokine Levels in Diagnosis and Management of Overactive Bladder in Children
Brief Title: Urinary Biomarkers in Overactive Bladder in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital Zagreb (Other)
Collaborators: University Hospital for Infectious Diseases, Croatia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: pOAB-CHZ-01
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Overactive Bladder
Keywords: Neurotrophins; Nerve Growth Factor; Brain-Derived Neurotrophic Factor; Urinary Biomarkers; Urodynamics; Anticholinergics; Children
MeSH Terms: conditions — Urinary Bladder, Overactive; Hereditary Sensory and Autonomic Neuropathies | interventions — oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other): Patients with overactive bladder will receive anticholinergic therapy: oral oxybutynin in daily dose 0.2-0.5 mg/kg divided in two daily doses for 3 to 6 months depending on treatment outcome assessed 3 months after start of intervention.
  Interventions: Drug: Oxybutynin

INTERVENTIONS:
Drug: Oxybutynin — Anticholinergic
  Other Names: Driptane

SUMMARY:
It is a single-center, prospective, interventional, single-arm study. Aim is to investigate which variables are significantly correlated with prolonged anticholinergic treatment (>6 months) in children with overactive bladder (OAB). Investigated variables will include urinary neurotrophins and inflammatory cytokines, sonographic biomarkers, symptom score scale, demographics, and urodynamic findings. Secondary aim is to analyze sensitivity and specificity of urinary biomarkers in diagnosis and management of OAB compared to urodynamics and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* urgency with or without frequency, incontinence, enuresis, or nocturia
* an unremarkable clinical examination
* a minimum of 3 micturitions per day
* informed oral and written consent from the child and both parents/legal guardian

Exclusion Criteria:

* acute urinary tract infection
* diseases of central or peripheral nerve system
* anomalies of lumbosacral region
* bladder outlet obstruction
* operative procedures or anomalies of urinary or genital tract
* hypercalcuria, diabetes mellitus, diabetes insipidus
* neurogenic bladder
* constipation or fecal incontinence
* urolithiasis, depression, eating disorders or cardio-metabolic diseases
* prior use of anticholinergic treatment during the last year

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Initial success | 6 months after start of intervention
  Nonresponse is defined as a 0% to 49% decrease, partial response is defined as a 50% to 89% decrease, response is defined as a 90% or greater decrease and full response is defined as a 100% decrease or less than 1 symptom occurrence monthly. Symptoms include urgency, daily incontinence, increased daytime frequency, enuresis, nocturia. Symptom frequency will be assessed using validated diary.

SECONDARY OUTCOMES:
Long-term success | 6 months after stop of intervention
  Relapse is defined as more than 1 symptom recurrence monthly, continued success is de-fined as no relapse in 6 months after the interruption of treatment.
Bladder wall thickness | 6 months after start of intervention
  Bladder wall thickness will be measured using ultrasonography.
Improvement in health-related quality of life measured by PedsQL 4.0 Generic Core questionnaire | 6 months after start of intervention
  Improvement is defined by increase in total and subscale scores by more than defined minimally clinical important difference for PedsQL 4.0 Generic Core questionnaire.
Urinary neurotrophins | 6 months after start of intervention
  Urine samples will be collected at urge sensation before and 6 months after start of intervention. Urinary nerve growth factor (NGF) and brain-derived neurotrophic factor (BDNF) levels normalized to urinary creatinine will be measured.
Urinary cytokines | 6 months after start of intervention
  Urine samples will be collected at urge sensation before and 6 months after start of intervention. Urinary inflammatory cytokines (MCP-1, MCP-2, MCP-3, CaCL-13) levels normalized to urinary creatinine will be measured.
Urodynamics | 6 months after start of intervention
  Urodynamic study will be investigated prior and 6 months after start of intervention. Maximum detrusor pressure will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Slaven Abdovic, MD, PhD, Principal Investigator — Children's Hospital Zagreb
Locations (1):
- Children's Hospital Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided